CLINICAL TRIAL: NCT03013985
Title: A Randomized Controlled Trial Comparing Glargine U300 and Glargine U100 for the Inpatient and Post-Hospital Discharge Management of Medicine and Surgery Patients With Type 2 Diabetes
Brief Title: Glargine U300 Hospital Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Guillermo Umpierrez, MD, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00091740
Record Dates: First submitted 2017-01-05; First posted 2017-01-09 (Estimated); Results first posted 2020-05-07 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-04

CONDITIONS: Type 2 Diabetes
Keywords: Blood glucose
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; insulin glulisine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Basal bolus insulin with glargine U300 and glulisine insulin (Experimental): Subjects treated with insulin prior to admission will receive 80% of the total daily dose (TDD) given as basal bolus insulin regimen with glargine U300 once daily plus rapid-acting glulisine insulin before meals. In insulin-naïve subjects treated with oral agents, the oral antidiabetic drugs will be discontinued and the bolus insulin dose described above will be given. Half of TDD will be given as glargine U300 and half as glulisine. To prevent hypoglycemia, if a subject is not able to eat, the dose of glulisine will be held.
  Interventions: Drug: Glargine U300; Drug: Glulisine Insulin
- Basal bolus insulin with glargine U100 and glulisine insulin (Active Comparator): Subjects treated with insulin prior to admission will receive 80% of the total daily dose (TDD) given as basal bolus insulin regimen with glargine U100 once daily plus rapid-acting glulisine insulin before meals. In insulin-naïve subjects treated with oral agents, the oral antidiabetic drugs will be discontinued and the bolus insulin dose as described above will be given. Half of TDD will be given as glargine U100 and half as glulisine. To prevent hypoglycemia, if a subject is not able to eat, the dose of glulisine will be held.
  Interventions: Drug: Glargine U100; Drug: Glulisine Insulin

INTERVENTIONS:
Drug: Glargine U300 — Glargine U300 is a new generation long-acting insulin.
  Other Names: Toujeo
  Arms: Basal bolus insulin with glargine U300 and glulisine insulin
Drug: Glargine U100 — Glargine U100 is a long-acting insulin.
  Other Names: Lantus
  Arms: Basal bolus insulin with glargine U100 and glulisine insulin
Drug: Glulisine Insulin — Glulisine is a mealtime insulin taken either 15 minutes before or 20 minutes after a meal.
  Other Names: Apidra

SUMMARY:
The purpose of this study is to find out if treatment with Glargine U300 when compared to Glargine U100 will result in similar sugar control in patients with Type 2 Diabetes (T2D), who are admitted to the hospital and then transition at home, after discharge from the hospital.

DETAILED DESCRIPTION:
Several randomized clinical trials done previously in medicine and surgical patients with T2D have shown that basal bolus regimen with glargine results in a lower mean daily blood glucose (BG) concentrations compared to the sole use of sliding scale regular insulin (SSI) and in lower rate of hospital complications. Glargine U300 results in similar improvement but in lower rate of hypoglycemia than treatment with glargine U100. No previous studies; however, have compared the efficacy and safety of glargine U300 in the management of hyperglycemia and diabetes in the hospital setting. This study will determine if treatment with glargine U300 has a similar glucose control in patients with diabetes admitted to the hospital and if glargine U300 will result in lower number of low blood sugars compared to glargine U100 .

ELIGIBILITY:
Inclusion Criteria:

* Males or females between > 18 years admitted to a general medicine or surgical service.
* Known histories of T2D treated with either diet alone, oral monotherapy, any combination of oral antidiabetic agents, short-acting GLP1-RA (exenatide, liraglutide) or insulin therapy with the exception of degludec and glargine U300.
* Subjects must have an admission/randomization BG > 140 mg and < 400 mg/dL without laboratory evidence of diabetic ketoacidosis (bicarbonate < 18 mEq/L, pH < 7.30, or positive serum or urinary ketones).

Exclusion Criteria:

* Subjects with increased BG concentration, but without a known history of diabetes.
* Patients treated with degludec or glargine U300, or with long-acting weekly GLP1-RA (weekly exenatide, dulaglutide or albiglutide).
* Patients with acute critical or surgical illness admitted to the ICU or expected to require admission to the ICU.
* Patients with clinically relevant hepatic disease (diagnosed liver cirrhosis and portal hypertension), corticosteroid therapy, or impaired renal function (eGFR< 30 ml/min).
* Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study.
* Female subjects who are pregnant or breast feeding at time of enrollment into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2019-03-22 (Actual); Study Completion 2019-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Umpierrez, MD, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pasquel FJ, Lansang MC, Khowaja A, Urrutia MA, Cardona S, Albury B, Galindo RJ, Fayfman M, Davis G, Migdal A, Vellanki P, Peng L, Umpierrez GE. A Randomized Controlled Trial Comparing Glargine U300 and Glargine U100 for the Inpatient Management of Medicine and Surgery Patients With Type 2 Diabetes: Glargine U300 Hospital Trial. Diabetes Care. 2020 Jun;43(6):1242-1248. doi: 10.2337/dc19-1940. Epub 2020 Apr 9. PMID 32273271

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 247 consented, 9 were not randomized, 27 failed to start (19 did not receive study medication, 1 had eGFR out of range, 7 had admission BG >400 mg/dl)
Period: Overall Study
Arm/Group | Basal Bolus Insulin With Glargine U300 and Glulisine Insulin | Basal Bolus Insulin With Glargine U100 and Glulisine Insulin
Started | 108 | 103
Completed | 92 | 84
Not Completed | 16 | 19
Not completed — Protocol Violation | 2 | 2
Not completed — Withdrawal by Subject | 14 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Basal Bolus Insulin With Glargine U300 and Glulisine Insulin | Basal Bolus Insulin With Glargine U100 and Glulisine Insulin | Total
Number analyzed (Participants) | 108 | 103 | 211
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (12.1) | 56.3 (12.4) | 56.7 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 39 | 85
  Male | 62 | 64 | 126
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 4 | 7
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 68 | 64 | 132
  White | 35 | 34 | 69
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 108 | 103 | 211

OUTCOME MEASURES:

1. Primary Outcome: Mean Daily Blood Glucose Concentration Inpatient
Description: The mean daily blood glucose concentration for all participants will be calculated by taking the average of all pre-meal and bedtime glucose values collected each day after the first day of therapy during the hospital stay.
Time Frame: up to 10 days (day of hospital discharge)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Basal Bolus Insulin With Glargine U300 and Glulisine Insulin | Basal Bolus Insulin With Glargine U100 and Glulisine Insulin
Number analyzed (Participants) | 92 | 84
mg/dL | 186 (40) | 184 (46)

2. Primary Outcome: Mean Daily Blood Glucose Concentration After Hospital Discharge
Description: Subjects will measure their blood sugar levels at home by finger stick before meals two or three times per day and record the readings in a diary. The readings will be averaged for each day and the mean daily blood glucose concentration will be calculated.
Time Frame: assessed from day 11 (day after hospital discharge) up to 3 months
Population: The outpatient has less number of participants compared to the in-hospital part due to a1c less tan required for outpatient part, participants not wanting to continue in the discharge part and/or admission to long term facilities where we were not able to administer study medication.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Basal Bolus Insulin With Glargine U300 and Glulisine Insulin | Basal Bolus Insulin With Glargine U100 and Glulisine Insulin
Number analyzed (Participants) | 41 | 45
mg/dL | 171.6 (44.8) | 164.5 (46.7)

3. Secondary Outcome: Mean Daily Glucose in Patients With Admission HbA1c Lower Than 8%
Description: Glycemic control will be measured by mean daily blood glucose concentration for subjects with HbA1c lower than 8% at admission. The average of all pre-meal and bedtime glucose values will be calculated.
Time Frame: up to 3 months post enrollment
Population: subjects with HbA1c lower than 8% at admission
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Basal Bolus Insulin With Glargine U300 and Glulisine Insulin | Basal Bolus Insulin With Glargine U100 and Glulisine Insulin
Number analyzed (Participants) | 27 | 31
mg/dL | 150 (14.4) | 134.4 (19.3)

4. Secondary Outcome: Mean Daily Glucose in Patients With Admission HbA1c Higher Than 8%
Description: Mean daily blood glucose concentration for subjects with HbA1c higher than 8% at admission will be recorded
Time Frame: up to 3 months post enrollment
Population: Patients with admission HbA1c higher than 8%
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Basal Bolus Insulin With Glargine U300 and Glulisine Insulin | Basal Bolus Insulin With Glargine U100 and Glulisine Insulin
Number analyzed (Participants) | 78 | 72
mg/dL | 152.3 (38.5) | 155.6 (36.5)

5. Secondary Outcome: Mean Daily Glucose in Patients With Length of Stay Shorter Than 3 Days
Description: Glycemic control will be conducted by measuring mean daily blood glucose concentration for subjects with length of hospital stay shorter than 3 days
Time Frame: Up to 3 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Basal Bolus Insulin With Glargine U300 and Glulisine Insulin | Basal Bolus Insulin With Glargine U100 and Glulisine Insulin
Number analyzed (Participants) | 92 | 84
mg/dL | 169.71 (42.35) | 196.72 (56.60)

6. Secondary Outcome: Mean Daily Glucose in Patients With Length of Stay Shorter Than 5 Days
Description: Glycemic control will be conducted by measuring mean daily blood glucose concentration for subjects with length of hospital stay shorter than 5 days
Time Frame: Up to 5 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Basal Bolus Insulin With Glargine U300 and Glulisine Insulin | Basal Bolus Insulin With Glargine U100 and Glulisine Insulin
Number analyzed (Participants) | 92 | 84
mg/dL | 193.53 (43.1) | 193.64 (42.6)

7. Secondary Outcome: Mean Daily Glucose in Patients With Length of Stay Longer Than 5 Days
Description: Glycemic control will be measured by mean daily blood glucose concentration for subjects with length of hospital stay longer than 5 days. The average of daily pre-meal and bedtime glucose values will be calculated.
Time Frame: Up to 10 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Basal Bolus Insulin With Glargine U300 and Glulisine Insulin | Basal Bolus Insulin With Glargine U100 and Glulisine Insulin
Number analyzed (Participants) | 92 | 84
mg/dL | 188.46 (34.7) | 174.55 (34.1)

8. Secondary Outcome: Percent of Blood Glucose 70-180 Measured by Point of Care Test
Description: Percent of Blood Glucose Readings in the 70-180 mg/dL Range Measured by Point of Care Test
Time Frame: 3 months post enrollment
Measure: Mean (Standard Deviation); unit: percentage of BG readings
Arm/Group | Basal Bolus Insulin With Glargine U300 and Glulisine Insulin | Basal Bolus Insulin With Glargine U100 and Glulisine Insulin
Number analyzed (Participants) | 92 | 84
percentage of BG readings | 50.3 (27.5) | 54.9 (29.3)

9. Secondary Outcome: Percent of Subjects With Hypoglycemic Events
Description: Percent of of subjects with hypoglycemic events (BG < 70 mg/dl) will be recorded.
Time Frame: 3 months post enrollment
Measure: Number; unit: percentage of subjects
Arm/Group | Basal Bolus Insulin With Glargine U300 and Glulisine Insulin | Basal Bolus Insulin With Glargine U100 and Glulisine Insulin
Number analyzed (Participants) | 92 | 84
percentage of subjects | 8.7 | 9.5

10. Secondary Outcome: Percent of Subjects With Severe Hypoglycemia
Description: Percent of subjects experiencing severe hypoglycemia (BG <54 mg/dl) will be recorded.
Time Frame: 3 months post enrollment
Measure: Number; unit: percentage of subjects
Arm/Group | Basal Bolus Insulin With Glargine U300 and Glulisine Insulin | Basal Bolus Insulin With Glargine U100 and Glulisine Insulin
Number analyzed (Participants) | 92 | 84
percentage of subjects | 0 | 6

11. Secondary Outcome: Number of Days of Hospital Stay
Description: The number of days of hospital stay for each subject will be recorded.
Time Frame: Up to 10 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Basal Bolus Insulin With Glargine U300 and Glulisine Insulin | Basal Bolus Insulin With Glargine U100 and Glulisine Insulin
Number analyzed (Participants) | 92 | 84
days | 6 [4 to 8] | 4 [3 to 7]

12. Secondary Outcome: Number Subjects With Cardiac Complications
Description: The number of subjects experiencing cardiac cardiac complications will be recorded.
Time Frame: 3 months post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Basal Bolus Insulin With Glargine U300 and Glulisine Insulin | Basal Bolus Insulin With Glargine U100 and Glulisine Insulin
Number analyzed (Participants) | 92 | 84
Participants | 5 | 11

13. Secondary Outcome: Number of Patients With Acute Renal Failure
Description: The number of subjects with a clinical diagnosis with documented new-onset abnormal renal function (increment in serum creatinine > 0.5 mg/dL from baseline).
Time Frame: 3 months post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Basal Bolus Insulin With Glargine U300 and Glulisine Insulin | Basal Bolus Insulin With Glargine U100 and Glulisine Insulin
Number analyzed (Participants) | 92 | 84
Participants | 1 | 1

14. Secondary Outcome: Hospital Mortality
Description: Number of hospital deaths that occur.
Time Frame: During hospital stay - up to 10 days
Measure: Number; unit: events
Arm/Group | Basal Bolus Insulin With Glargine U300 and Glulisine Insulin | Basal Bolus Insulin With Glargine U100 and Glulisine Insulin
Number analyzed (Participants) | 92 | 84
events | 0 | 2

ADVERSE EVENTS:
Time Frame: 3 months.
Arm/Group | Basal Bolus Insulin With Glargine U300 and Glulisine Insulin | Basal Bolus Insulin With Glargine U100 and Glulisine Insulin
All-Cause Mortality (participants affected / at risk) | 0/108 | 2/103
Serious Adverse Events (participants affected / at risk) | 21/108 | 21/103
Other Adverse Events (participants affected / at risk) | 10/108 | 18/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Basal Bolus Insulin With Glargine U300 and Glulisine Insulin (N=108) | Basal Bolus Insulin With Glargine U100 and Glulisine Insulin (N=103)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 3 (3)
Gastroentestinal disorder (Gastrointestinal disorders) | 4 (6) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Chronic Heart Failure (Cardiac disorders) | 4 (6) | 8 (10)
Infection (General disorders) | 3 (4) | 4 (4)
Surgery (General disorders) | 2 (2) | 0 (0)
Stroke (Vascular disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Malfunctioning Peripherally Inserted Central Catheter (Surgical and medical procedures) | 1 (1) | 1 (1)
Syncope (Cardiac disorders) | 1 (1) | 0 (0)
Skin graft failure (Immune system disorders) | 0 (0) | 1 (1)
Numbness on right side of body (Nervous system disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ICU admission (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Basal Bolus Insulin With Glargine U300 and Glulisine Insulin (N=108) | Basal Bolus Insulin With Glargine U100 and Glulisine Insulin (N=103)
Gastroparesis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Hyperglycemia (Endocrine disorders) | 0 (0) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Infection (General disorders) | 0 (0) | 3 (3)
Leg Swelling (General disorders) | 0 (0) | 2 (3)
Pain (General disorders) | 1 (1) | 2 (3)
Polysubstance abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Skin Graft revision (Surgical and medical procedures) | 0 (0) | 1 (1)
Scrotal Bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Social (homelessness) (Social circumstances) | 0 (0) | 1 (1)
Trauma (General disorders) | 4 (4) | 1 (1)
Tremors (General disorders) | 1 (1) | 0 (0)
Wound Check (Surgical and medical procedures) | 1 (1) | 1 (1)
Cerumen Impaction (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-28): https://cdn.clinicaltrials.gov/large-docs/85/NCT03013985/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-28): https://cdn.clinicaltrials.gov/large-docs/85/NCT03013985/ICF_001.pdf